CLINICAL TRIAL: NCT00730236
Title: A Phase III Study of Microsomal Triglyceride Transfer Protein (MTP) Inhibitor AEGR-733 in Patients With Homozygous Familial Hypercholesterolemia on Current Lipid-lowering Therapy
Brief Title: A Safety and Efficacy Study of AEGR-733 to Treat Homozygous Familial Hypercholesterolemia (FH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEGR-733-005 / UP1002; NCT00603161 (obsolete NCT alias)
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2013-01

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AEGR-733 (Experimental)
  Interventions: Drug: AEGR-733

INTERVENTIONS:
Drug: AEGR-733 — 5-80 mg daily by mouth for 1.5 yrs
  Other Names: lomitapide; BMS-201038

SUMMARY:
The goal of this trial is to study the effects of AEGR-733 on LDL cholesterol, other lipids as well as measures of safety over the long-term.

DETAILED DESCRIPTION:
Homozygous familial hypercholesterolemia (FH) is a serious life-threatening genetic disease. Total plasma cholesterol levels are generally over 500 mg/dl and markedly premature cardiovascular disease is the major consequence. Untreated, most patients develop atherosclerosis before age 20 and generally do not survive past age 30. The primary goal of therapy involves reducing cholesterol (specifically, LDL cholesterol) and preventing coronary artery disease. Unfortunately, patients with homozygous FH are minimally responsive or unresponsive to available drug therapy and thus there are limited treatment options. The current standard of care is LDL apheresis, a physical method of removing the plasma of LDL cholesterol which can transiently reduce cholesterol by more than 50%. However, there is rapid re-accumulation of LDL cholesterol in plasma, and therefore apheresis has to be repeated frequently (every 1-2 weeks) and requires 2 separate sites for IV access. Although anecdotally this procedure may delay the onset of atherosclerosis, it is laborious, expensive, and not readily available. Furthermore, although it is a procedure that is generally well tolerated, the fact that it needs frequent repetition and IV access can be challenging for many of these young patients. Therefore, there is a tremendous unmet medical need for new medical therapies for this orphan disease.

AEGR-733 is a novel oral therapeutic agent for hypercholesterolemia. Its mechanism involves inhibition of microsomal triglyceride transfer protein, resulting in a reduction of LDL cholesterol. Earlier studies in patients with homozygous FH reveal AEGR-733 is highly effective in lowering LDL cholesterol, yet long term safety and efficacy need to be established.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age
2. Diagnosis of functional homozygous FH by at least one (a-c) of the following clinical criteria:

   * documented functional mutation(s) in both LDL receptor alleles or alleles known to affect LDL receptor functionality OR
   * skin fibroblast LDL receptor activity less than 20% normal OR
   * untreated TC greater than 500 mg/dL AND TG less then 300 mg/dL AND both parents have documented TC greater than 250 mg/dL
3. Concurrent lipid lowering medication/apheresis must be stable for at least 6 weeks before the baseline visit and must remain stable for the first 26 weeks.
4. Body weight at least 40 kg and less than 136 kg
5. Negative screening pregnancy test if female of child-bearing potential (females of child-bearing potential and all males must be following a medically accepted form of contraception)
6. Subjects must be willing to comply with all study-related procedures

Exclusion Criteria:

1. Uncontrolled hypertension
2. History of chronic renal insufficiency
3. History of biopsy proven cirrhosis or abnormal LFTs at screening (AST or ALT greater than 2 x upper limit of normal and/or Total Bilirubin greater than or equal to 1.5 mg/dl unless patient has unconjugated hyperbilirubinemia due to Gilbert's syndrome)
4. Chronic hepatitis B or chronic hepatitis C
5. Any major surgical procedure occurring less than 3 months prior to the screening visit
6. Cardiac insufficiency defined by the NYHA classification as functional Class III or Class IV
7. Previous organ transplantation
8. History of a non-skin malignancy within the previous 3 years
9. Male subjects reporting more than 2 drinks per day or females reporting more than 1 drink per day (1 drink= 12 oz beer, 1 oz hard liquor, 5 oz wine).
10. Participation in an investigational drug study within 6 weeks prior to the screening visit
11. Known significant gastrointestinal bowel disease or malabsorption such as inflammatory bowel disease or chronic pancreatitis requiring use of daily pancreatic enzymes.
12. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
13. Certain prohibited medications known to be potentially hepatotoxic, especially those that can induce microvesicular or macrovesicular steatosis. These include but are not limited to: accutane, amiodarone, heavy acetaminophen use (4g/day greater than 3 x q week), methotrexate, tetracyclines,and tamoxifen
14. Documented diagnosis of any of the following pulmonary conditions: Asthma, Chronic Obstructive Pulmonary Disease (COPD), Idiopathic pulmonary fibrosis
15. Documented diagnosis of any of the following liver diseases: Nonalcoholic Steatohepatitis, Alcoholic liver disease, Autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, hemochromatosis, alpha 1 anti-trypsin deficiency.
16. Current use of corticosteroids or betaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sumeray, MD, Study Director — Aegerion Pharmaceuticals, Inc.; Marina Cuchel, MD, PhD, Principal Investigator — Univerity of Pennsylvania
Locations (10):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (2):
  - Robarts Research Institute, London, Ontario
  - Lipid Clinic and University of Montreal Community Genomic Medicine Center, Chicoutimi, Quebec
- Italy (4):
  - Dipartimento di Medicina Clinica e Della Patalogie Emergenti, Palermo, Sicily
  - Medicina Interna Universitaria, Ferrara
  - Centro Universitario Dislipidemie, Milan
  - Dipartimento di Clinica e Terapia Medica, Roma
- South Africa (2):
  - Cardiology Research, Bloemfontein
  - University of Capetown, Cape Town

REFERENCES:
- [Background] Cuchel M, Bloedon LT, Szapary PO, Kolansky DM, Wolfe ML, Sarkis A, Millar JS, Ikewaki K, Siegelman ES, Gregg RE, Rader DJ. Inhibition of microsomal triglyceride transfer protein in familial hypercholesterolemia. N Engl J Med. 2007 Jan 11;356(2):148-56. doi: 10.1056/NEJMoa061189. PMID 17215532
- [Result] Cuchel M, Meagher E, Marais AD, et.al. Abstract 1077: A phase III study of microsomal triglyceride transfer protein inhibitor lomitapide (AEGR-733) in patients with homozygous familial hypercholesterolemia: interim results at 6 months. Circulation, Nov 2009; 120: S441
- [Derived] Larrey D, D'Erasmo L, O'Brien S, Arca M; Italian Working Group on Lomitapide. Long-term hepatic safety of lomitapide in homozygous familial hypercholesterolaemia. Liver Int. 2023 Feb;43(2):413-423. doi: 10.1111/liv.15497. Epub 2022 Dec 30. PMID 36520008
- [Derived] Averna M, Cefalu AB, Stefanutti C, Di Giacomo S, Sirtori CR, Vigna G. Individual analysis of patients with HoFH participating in a phase 3 trial with lomitapide: The Italian cohort. Nutr Metab Cardiovasc Dis. 2016 Jan;26(1):36-44. doi: 10.1016/j.numecd.2015.11.001. Epub 2015 Nov 11. PMID 26723464
- [Derived] Stefanutti C, Blom DJ, Averna MR, Meagher EA, Theron Hd, Marais AD, Hegele RA, Sirtori CR, Shah PK, Gaudet D, Vigna GB, Sachais BS, Di Giacomo S, du Plessis AM, Bloedon LT, Balser J, Rader DJ, Cuchel M; Phase 3 HoFH Lomitapide Study Investigators. The lipid-lowering effects of lomitapide are unaffected by adjunctive apheresis in patients with homozygous familial hypercholesterolaemia - a post-hoc analysis of a Phase 3, single-arm, open-label trial. Atherosclerosis. 2015 Jun;240(2):408-14. doi: 10.1016/j.atherosclerosis.2015.03.014. Epub 2015 Mar 14. PMID 25897792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed from 18 Dec 2007 to 13 Oct 2011. A total of 11 medical clinics participated in the study.
Pre-assignment Details: 6-week Run-in Phase. Following screening, patients entered a 6-week Run-in Phase to stabilize their regimen of current lipid-lowering therapy(ies) and to be placed on a low-fat diet containing <20% energy from fat.
Groups:
- Lomitapide Escalated: Lomitapide escalated with an initial oral dose of 5 mg/day for 2 weeks and then escalated at 4 week intervals to 60 mg/day. In rare situations (1 patient)who met strict safety and efficacy criteria could have their dose escalated to 80 mg/day.
Period: Overall Study
Arm/Group | Lomitapide Escalated
Started | 29
Completed | 23
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7
  Canada | 5
  South Africa | 11
  Italy | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Percent change from Baseline in LDL-C
Time Frame: Baseline and Week 26
Population: Intention To Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Change | -40.1 (31.25)

2. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC)
Description: Percent change from Baseline in TC
Time Frame: Baseline and Week 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Change | -36.4 (28.2)

3. Secondary Outcome: Percent Change From Baseline for Apolipoprotein B (Apo B)
Description: Percent change from Baseline for Apo B
Time Frame: Baseline and Week 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Change | -39.4 (30.01)

4. Secondary Outcome: Percent Change From Baseline in Triglycerides
Description: Percent change from Baseline in triglycerides
Time Frame: Baseline and Week 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Change | -29.0 (55.72)

5. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change from Baseline in HDL-C
Time Frame: Baseline and Week 26
Population: ITT Population
Measure: Median (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Change | -6.9 (19.76)

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C
Description: Percent change from Baseline in non-HDL-C
Time Frame: Baseline and Week 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Change | -40.0 (29.66)

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein AI (Apo AI)
Description: Percent change from Baseline in Apo AI
Time Frame: Baseline and Week 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Change | -6.5 (16.12)

8. Secondary Outcome: Absolute Change From Baseline in Hepatic Fat Percent
Description: Absolute change from Baseline in hepatic fat percent
Time Frame: Baseline and Week 78
Population: All patients treated
Measure: Mean (Standard Deviation); unit: Percent Hepatic Fat
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
Percent Hepatic Fat | 6.9 (5.03)

9. Secondary Outcome: Absolute Change From Baseline in Alanine Aminotransferase (ALT)
Description: Absolute change from Baseline in ALT
Time Frame: Baseline and Week 78
Population: All patients treated
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
U/L | 15.0 (29.05)

10. Secondary Outcome: Absolute Change From Baseline in Aspartate Aminotransferase (AST)
Description: Absolute change from Baseline in AST
Time Frame: Baseline and Week 78
Population: All patients treated
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
U/L | 8.9 (20.22)

11. Secondary Outcome: Absolute Change From Baseline in Total Bilirubin
Description: Absolute change from Baseline in total bilirubin
Time Frame: Baseline and Week 78
Population: All patients treated
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
mg/dL | 0.1 (0.30)

12. Secondary Outcome: Absolute Change From Baseline in Weight
Description: Absolute change from Baseline in weight
Time Frame: Baseline and Week 78
Population: All patients treated
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 29
kg | -2.3 (3.46)

ADVERSE EVENTS:
Time Frame: First dose to 28 days post treatment
Arm/Group | Lomitapide Escalated
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lomitapide Escalated (N=29)
Angina pectoris (Cardiac disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Coronary artery arteriosclerosis (Cardiac disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lomitapide Escalated (N=29)
Diarrhoea (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 10
Abdominal discomfort (Gastrointestinal disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 5
Chest pain (General disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 5
Constipation (Gastrointestinal disorders) | 6
Weight decreased (Investigations) | 7
Headache (Nervous system disorders) | 3
Flatulence (Gastrointestinal disorders) | 6
Influenza (Infections and infestations) | 6
Aspartate aminotransferase increased (Investigations) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 5
Nasopharyngitis (Infections and infestations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dizziness (Nervous system disorders) | 3
Gastroenteritis (Infections and infestations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Hot flush (Vascular disorders) | 2
Palpitations (Cardiac disorders) | 3
Rectal tenesmus (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Conjunctivitis (Eye disorders) | 2
Defaecation urgency (Gastrointestinal disorders) | 2
Eructation (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Gingivitis (Gastrointestinal disorders) | 2
Hepatic steatosis (Hepatobiliary disorders) | 2
Bronchitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 2
Transaminases increased (Investigations) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The CTAs generally envision a multisite publication, with the PI's right to publish individually if the pooled publication does not occur within 12 months of study completion. Sponsor has a 45 to 60 day review/approval period to request deletion of confidential information or to request limited deferral to protect its proprietary technology. In one case, the publication provision is more general, specifying that the Sponsor and clinical site will agree on the manner/terms of publication.